CLINICAL TRIAL: NCT00211042
Title: Observational, Multicenter Study of Subjects With Pure Red Cell Aplasia Associated With r-HuEPO Treatment
Brief Title: A Study of Patients With Pure Red Cell Aplasia Associated With Recombinant Human Erythropoietin Treatment
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004393; EPO-IMU-301 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Pure Red-cell Aplasia
Keywords: Pure red-cell aplasia; Anemia; Red blood cells; Epoetin alfa (Eprex); Anti-erythropoietin antibodies; Recombinant human erythropoietin
MeSH Terms: conditions — Red-Cell Aplasia, Pure; Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pure Red Cell Aplasia (PRCA): This study will examine the relationship of the presence of anti-erythropoietin antibodies to the clinical course and outcome of participants currently or previously treated with recombinant human erythropoietin and who have PRCA identified from all notified reports (spontaneous postmarketing reports or from clinical trials reports).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. No medication will be given to the participants. Participants will receive standard-of-care treatment from their individual physicians.

SUMMARY:
The purpose of this study is to investigate the relationship of anti-erythropoietin antibodies to the clinical course and outcome of pure red cell aplasia (PRCA) in participants currently or previously treated with recombinant human erythropoietin.

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), observational (study in which the investigators/physicians observe the participant's data and measure their outcomes) study. Approximately 150 participants will be enrolled in this study. The study consists of an initial observation phase and extended observation period. An initial observation phase starting at enrollment and ending when 24 months have elapsed since the date of loss of efficacy (LOE), supplemented with retrospective data collection for the period between LOE date and date of enrollment in the study. Participants remaining epoetin alfa (EPO-Ab) positive 24 months after LOE will enter a 2-year extended observation period. Study visits will take place every month during the initial observation phase and data will be collected every 6 months during the extended observation phase. Safety evaluations will include assessment of adverse events, clinical laboratory tests, vital signs, and physical examination which will be monitored throughout the study. The total study duration for each participant will be approximately for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Pure red cell aplasia (PRCA) associated with recombinant human erythropoietin (r-HuEPO) treatment
* Anemia unresponsive to r-HuEPO treatment
* PRCA associated with erythropoietin treatment followed by a sudden decrease (more than or equal to 2 gram per deciliter within 30 days) in a previously stable hemoglobin level

Exclusion criteria:

- Participants who are not fulfilling the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with Pure Red Cell Aplasia (PRCA)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2004-02; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Pure Red Cell Aplasia (PRCA) outcome (Initial observation phase) | Up to 24 months after the date of loss of efficacy
  The PRCA outcome is measured by anti-epoetin alfa qualitative test. Persistence of PRCA is defined as: 1) absolute reticulocyte count less than 30,000 per cubic millimeter; and/or 2) no reversal of erythroblastopenia on repeated bone marrow testing. Resolution of PRCA is defined as: 1) absolute reticulocyte count greater than or equal to 30,000 per cubic millimeter; and/or 2) reversal of erythroblastopenia on repeated bone marrow testing.
Number of participants with pure red cell aplasia outcome (Extended observation phase) | Up to 2 years after the enrollment in the extended observation phase
  Participants remaining anti-epoetin alfa positive 24 months after loss of efficacy will enter in the extended observation period.
Overall clinical outcome of pure red cell aplasia (Initial observation phase) | Up to 24 months after the date of loss of efficacy
  The overall clinical outcome is evaluated by anti-epoetin alfa qualitative test. Overall clinical status will be recorded at each visit in the initial and extended observation phases using a categorical scale (improved, same, worsened, death). In case of death, the date and cause of death along with the the date and cause of death will be recorded.
Overall clinical outcome of pure red cell aplasia (Extended observation phase) | Up to 2 years after the enrollment in the extended observation phase

SECONDARY OUTCOMES:
Different treatment modalities with pure red cell aplasia outcome (Initial observation phase) | Up to 24 months after the date of loss of efficacy
Different treatment modalities with pure red cell aplasia outcome (Extended observation phase) | Up to 2 years after the enrollment in the extended observation phase
Risk factors for Loss of Efficacy (LOE) and pure red cell aplasia (PRCA) outcome | Period between LOE date and date of enrollment in the study
  This data will be collected retrospectively and the date of LOE will be determined by the sponsor based upon reported data. PRCA duration groups will be summarized by potential risk factors to evaluate the relationship of risk factors to the duration of PRCA.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L. L. C. Clinical trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (21):
- Brazil (2):
  - Santos
  - São Paulo
- Saskatoon, Saskatchewan, Canada
- Germany (2):
  - Darmstadt
  - Hannoversch Münden
- Tvnsberg, Norway
- Bloemfontein, South Africa
- Sweden (4):
  - Karlshamn
  - Linköping
  - Stockholm
  - Trollhättan
- N/a N/a, Thailand
- United Kingdom (9):
  - Birmingham
  - Chelmsford
  - Edinburgh
  - London
  - Manchester
  - Santander N/A
  - Telford
  - Valencia
  - Westcliff-on-Sea